CLINICAL TRIAL: NCT05421052
Title: Unmet Health Needs Among Sohag University Students
Brief Title: Unmet Health Needs Among Students
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mariam Mohamed Ahmed, Demonstrator at public health and community medicine department, Sohag University
Other Study IDs: Soh-med-22-06-04
Record Dates: First submitted 2022-06-12; First posted 2022-06-16 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Unmet Health Needs

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Unmet health needs — The students who have unmet health needs during the last 6 months will respond to the questionnaire to assess the causes and other factors

SUMMARY:
The concept of unmet health needs refers to the difference between health services thought necessary to treat a particular health problem and services actually received. A person who perceived the need to receive medical services but who has not obtained these services has unmet health care needs. Unmet health care may result from limited availability or unavailability of health care services, when or where they were required. Also it can be caused from individual accessibility problem, such as cost or transportation, or from acceptability problem, such as attitude toward and knowledge about health care.so, the investigators will assess the unmet health needs and identify the causes.

ELIGIBILITY:
Inclusion Criteria:

* all students who are more than 18 years old and approve to participate in the study

Exclusion Criteria:

* any students who refuse to participate in the study or who are under 18 years old

Ages: 18 Years to 35 Years | Sex: All
Age Groups: Adult
Study Population: Sohag university students from both sexes above 18 years old from ( faculty medicine, pharmacy, education, specific education )
Sampling Method: Probability Sample
Enrollment: 415 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of the unmet health needs of Sohag university students. | Assess the unmet health needs of the students during the last 6 months
  Identify the most important causes of unmet health needs among students by answering the questionnaire

SECONDARY OUTCOMES:
Assessment of the students' awareness and attitude towards Sohag University Medical Center | Assess the students' use of the University Medical Center during the last year
  The students will answer the questionnaire to know if they know about the University Medical Center or not and how the evaluate it.